CLINICAL TRIAL: NCT04469686
Title: 3-Arm Randomized Placebo Controlled Double Blind Phase 3 Study to Evaluate Safety and Efficacy of Once-Daily and Twice-Daily Hydrocortisone Acetate 90 mg Suppository Administered With a Sephure Applicator in Subjects With Ulcerative Colitis
Brief Title: Phase 3 Study to Evaluate the Safety and Efficacy of Hydrocortisone Acetate Suppositories
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cristcot LLC (Industry)
Collaborators: Cristcot HCA LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS1221; 2019-003596-19 (EudraCT Number)
Record Dates: First submitted 2020-07-02; First posted 2020-07-14 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Proctitis
MeSH Terms: interventions — hydrocortisone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Twice Daily - Active (Experimental): Twice daily 90 mg hydrocortisone acetate suppository administered with Sephure suppository applicator
  Interventions: Combination Product: Twice daily 90 mg hydrocortisone acetate suppository administered with Sephure applicator
- Once Daily - Active (Experimental): Once daily 90 mg hydrocortisone acetate and once daily placebo suppository administered with Sephure suppository applicator
  Interventions: Combination Product: Once daily 90 mg hydrocortisone acetate or placebo suppository administered with Sephure applicator
- Placebo (Placebo Comparator): Twice daily placebo suppository administered with Sephure suppository applicator
  Interventions: Combination Product: Twice daily placebo suppository administered with Sephure applicator

INTERVENTIONS:
Combination Product: Twice daily 90 mg hydrocortisone acetate suppository administered with Sephure applicator — Twice daily 90 mg hydrocortisone acetate suppository administered with Sephure applicator
  Other Names: Twice Daily - Active
  Arms: Twice Daily - Active
Combination Product: Once daily 90 mg hydrocortisone acetate or placebo suppository administered with Sephure applicator — Once daily 90 mg hydrocortisone acetate or placebo suppository administered with Sephure applicator
  Other Names: Once Daily - Active
  Arms: Once Daily - Active
Combination Product: Twice daily placebo suppository administered with Sephure applicator — Twice daily placebo suppository administered with Sephure applicator
  Other Names: Twice Daily - Placebo
  Arms: Placebo

SUMMARY:
A randomized, multi-center, double-blind, three arm placebo-controlled study in male and non-pregnant, non-lactating female subjects aged 18 years to examine the safety and efficacy of two dosing regimens of hydrocortisone acetate 90 mg suppository administered with the Sephure applicator for the treatment of ulcerative colitis of the rectum.

DETAILED DESCRIPTION:
Hydrocortisone acetate 90 mg or placebo will be administered as a rectal suppository with a Sephure suppository applicator. Two arms of the study will receive different dosage regimens of hydrocortisone acetate, and the third arm will receive placebo. All subjects will administer the study drug twice a day; once in the morning and once in the evening for 28 days.

The study population will consist of male and non pregnant, non lactating females aged 18 years and older with a confirmed diagnosis of active UC of the rectum.

ELIGIBILITY:
Inclusion Criteria:

* Male or non pregnant, non lactating females aged 18 years and older.
* Subjects with a confirmed diagnosis of active UC of the rectum, extending no more than 15 centimeters (cm) (5.9 inches) proximal to the anal verge as assessed by colonoscopy performed at Visit 2. Note: Subjects may have a history of more extensive UC (e.g., pancolitis), but have active disease only in the rectum at the time of enrollment.
* Modified Mayo sub score for stool frequency of 1 3.
* Modified Mayo sub score for rectal bleeding of 0 2.
* Modified Mayo endoscopic sub score of 2 3.
* Total Modified Mayo Score (without physician global assessment) of 4-8.

Exclusion Criteria:

* History or current diagnosis of bacterial or other infectious colitis, radiation enteritis and radiation proctitis, Crohn's disease, collagenous colitis and indeterminate colitis.
* Prior gastrointestinal surgery except appendectomy, cholecystectomy, and hernia.
* Concomitant active lower gastrointestinal disease (except Irritable Bowel Syndrome) or distortion of intestinal anatomy.
* Bleeding hemorrhoids at the time of enrollment.
* Acute diverticulitis at the time of enrollment.
* Acute or chronic pancreatitis at the time of enrollment.
* Unmanaged celiac disease at the time of enrollment.
* Positive stool test for enteric pathogens, Clostridium difficile, or presence of ova and parasites.
* Taking a prohibited medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Clinical remission measured using the Modified Mayo Score | 28 days
  To evaluate the the efficacy of two dosage regimens of the study drug

SECONDARY OUTCOMES:
Reduction of stool frequency measured using Mayo Scoring sub score of stool frequency | 28 days
  To assess the change in stool frequency
Rectal bleeding measured using Mayo Scoring sub-score of rectal bleeding equal to 0 | 28 days
  To assess the change in rectal bleeding

OTHER OUTCOMES:
Quality of Life assessed measured using IBDQ validated questionnaire | 28 days
  To examine the quality of life of patients
Grading of disease severity measure using Mayo Scoring sub-score of Physician's Global Assessment | 28 days
  To assess disease severity
Concentrations of hydrocortisone acetate using pharmacokinetic sampling | 28 days
  To evaluate the exposure of hydrocortisone acetate levels for safety

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Davagian, Study Director — Cristcot LLC
Locations (189):
- United States (51):
  - Clinical Research Associates LLC, Huntsville, Alabama
  - Om Research, Apple Valley, California
  - Om Research, Camarillo, California
  - Precision Research, El Cajon, California
  - Om Research, Lancaster, California
  - Southern CA Research Institute Medical Group/W Gastroenterology Medical Group, Los Angeles, California
  - Cornell Medical Research, Newport Beach, California
  - California Medical Research Associates Inc, Northridge, California
  - Clinical Applications Laboratories Inc, San Diego, California
  - I.H.S. Health, LLC, Kissimmee, Florida
  - Homestead Associates in Research, Miami, Florida
  - Rejuvaline Medical Research, Miami, Florida
  - Ezy Medical Research, Co., Miami, Florida
  - US Associates In Research, Miami, Florida
  - Gastro Health Research of Miami, Miami, Florida
  - GI PROS Research, Naples, Florida
  - Gastroenterology of Greater Orlando, Orange City, Florida
  - Revival Clinical Research, Orlando, Florida
  - BRCR Global Clinical Research, Plantation, Florida
  - International Center for Research, Tampa, Florida
  - One Health Research Clinic Atlanta, Johns Creek, Georgia
  - Comprehensive Gastrointestinal Health, LLC, Northbrook, Illinois
  - Cedar Valley Medical Specialists, P.C., Waterloo, Iowa
  - Combined Gastro LLC, Lafayette, Louisiana
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Revive Research Institute, Farmington Hills, Michigan
  - Clinical Research Institute of Michigan, Troy, Michigan
  - Sanmora Bespoke Clinical Research Solutions, LLC., East Orange, New Jersey
  - Westchester Putnam Gastro, Carmel, New York
  - Peters Medical Research, High Point, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Gastro Health Research, Cincinnati, Ohio
  - NexGen Research, Lima, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Gastroenterology Associates, Greenville, South Carolina
  - Gastro Associates of Greenville, Greenville, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - Allied Digestive Disease Center, Cypress, Texas
  - Dr. Mouhamad R. Al-Sabbagh, Houston, Texas
  - Elixir Research Group, Houston, Texas
  - Digestive Health Associates, Houston, Texas
  - Aspira International, Pasadena, Texas
  - LINQ Research LLC, Pearland, Texas
  - Southern Star Research Institute, LLC., San Antonio, Texas
  - Medrasa Clinical, Sherman, Texas
  - Spring Gastroenterology Associates, Spring, Texas
  - Texas Gastroenterology Associates, Spring, Texas
  - Velocity Clinical Research/Gut Whisperer, West Jordan, Utah
- Bulgaria (6):
  - Hospital Sveti Panteleimon, Plovdiv
  - Medical Center Hipokrat - H, Plovdiv
  - LTD Diagnostic Consultative Center 1, Sliven
  - Medical Center Excelsior 2, Sofia
  - Medical Center Excelsior, Sofia
  - University Hospital Tsaritsa Yoanna-ISUL, Sofia
- China (4):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Humanity & Health Clinical Trial Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Hvidovre Hospital, Hvidovre
  - Zealand University Hospital, Koge, Køge
- France (6):
  - CHU Lille - Hôpital Claude Huriez, Lille, Cedex
  - CHU TOURS. Service d'hépato-Gastro-entérologie, Chambray-lès-Tours
  - CHU Montpellier - Hopital Saint Eloi, Montpellier
  - Hôpital Lyon Sud - HCL, Pierre-Bénite
  - CHU de Saint-Étienne, Saint-Priest-en-Jarez
  - Hopital Rangueil, Toulouse
- Georgia (4):
  - JSC,, Vian", Kutaisi
  - LTD "Aversi Clinic", Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
  - LTD "Multi-Profile Clinic Consilium Medulla", Tbilisi
- Germany (5):
  - Praxis Dr. Michael R. Mross, Berlin
  - Studiengesellschaft BSF UG, Halle
  - EuGastro GmbH, Leipzig
  - Gastro Campus Research GbR, Münster
  - Zentrum für Gastroenterologie Saar MVZ GmbH, Saarbrücken
- India (13):
  - Ahmedabad Bariatrics & Cosmetics Private Limited (Asian Bariatrics), Ahmedabad, Gujarat
  - ICON Hospital, Ahmedabad, Gujarat
  - Sanjivani Superspeciality Hospital, Ahmedabad, Gujarat
  - Gujarat Gastro and Vascular Hospital, Surat, Gujarat
  - Lokmanya Tilak Municipal Medical College & Lokmanya Tilak Municipal General Hospital, Mumbai, Maharashtra
  - Midas Institute of Gastroenterology, Nagpur, Maharashtra
  - B.J. Government Medical College and Sassoon General Hospital, Pune, Maharashtra
  - Ashwin Medical Foundation Multispeciality Hospital, Pune, Maharashtra
  - Acharya Vinoba Bhave Rural Hospital, Wardha, Maharashtra
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - SIMS Hospital, Chennai, Tamil Nadu
  - Sir Ganga Ram Hospital,, Delhi
  - Pushpawati Singhania Research Institute, New Delhi
- Italy (5):
  - Università di Cagliari, Dipartimento di Scienze mediche e sanità pubblica, Monserrato, Cagliari
  - Ospedale: Azienda Policlinico Universitario Bari, Bari
  - Università della Campania "Luigi Vanvitelli", Napoli
  - Ospedale di Padova, Padua
  - A.O. Ordine Mauriziano di Torino, Torino
- Jordan (7):
  - Al Khalidi Hospital and Medical Center, Amman
  - Istishari Hospital, Amman
  - The Specialty Hospital Advanced Clinical Center, Amman
  - Istiklal Hospital, Amman
  - Jordan University Hospital, Amman
  - Irbid Specialty Hospital/Clinical Research Center, Irbid
  - Pharmaceutical Research Center/Jordan University of Science and Technology, Irbid
- Lebanon (3):
  - Saint George Hospital University Medical Center, Beirut
  - Dr. Bilal Hotayt Gastroenterology, Beirut
  - Hammoud Hospital University Medical Center, Sidon
- Nini Hospital, Tripoli, Libya
- Moldova (2):
  - Institutul de Cardiologie Consultative Department, RTL Clinic, Chisinau
  - Republican Hospital "Timofei Moșneaga", Consultative Department, Policlinic, Chisinau
- Philippines (10):
  - Cebu Doctors' University Hospital, Cebu City
  - The Medical City Iloilo, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - The Medical City Clark, Mabalacat
  - Makati Medical Center, Makati City
  - Manila Doctors Hospital, Manila
  - The Medical City Ortigas, Pasig
  - National Kidney and Transplant Institute, Quezon City
  - St. Luke's Medical Center, Quezon City
  - Cardinal Santos Medical Center (CSMC), San Juan City
- Poland (15):
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Uromed Jakub Koteras Twoja Przychodnia- Szczecińskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Vitamed Galaj i Cichomski Sp.j., Bydgoszcz
  - Osrodek Badan Klinicznych CLINSANTE S.C. Ewa Galczak-Nowak, Malgorzata Trzaska, Bydgoszcz
  - Centrum Medyczne Lukamed Joanna Luka Wendrowska, Chojnice
  - Centrum Medyczne MBB-MED, Chrzanów
  - Centrum Medyczne CLW-MED Aneta Cichomska, Joanna Luka-Wendrowska, Grudziądz
  - Karkonoskie Centrum Badan Klinicznych Lexmedica Sp. z o.o, Jelenia Góra
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - AMICARE Sp. z o.o. sp. k., Lodz
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Sonomed Sp. z o.o., Szczecin
  - Medical Concierge Centrum Medyczne, Warsaw
  - Medical Network Spółka z o.o., Warsaw
  - Melita Medical Centrum Medyczne, Wroclaw
- Romania (8):
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic 'Dr Ion Cantacuzino', Bucharest
  - Clinical Institute Fundeni, Gastro Enterology Department No.2, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Regional Institute of Gastroenterology and Hepatology "Prof. Dr. Octavian Fodor" Cluj-Napoca, Cluj-Napoca
  - Gastromedical SRL, Iași
  - Tirgu-Mures Country Clinical Hospital, Târgu Mureş
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Russia (7):
  - SBI of HE "Ryazan State Medical University n.a. ac. I.P. Pavlov" of the MoH of the RF on the base of the SBI of the Ryazan Region "Regional Clinical Hospital", Ryazan
  - Federal State Budgetary Military Educational Institution of Higher Education "Military and Medical Academy named after S.M. Kirov" of the Ministry of Defence of the Russian Federation; 2nd Therapy Chair for Advanced Training of Physicians, Saint Petersburg
  - Federal State Budgetary Military Educational Institution of Higher Education "Military and Medical Academy named after S.M. Kirov" of the Ministry of Defense of the Russian Federation; Chair and Clinic of Hospital Therapy n. a. Professor V.N. Sirotinin, Saint Petersburg
  - LLC 'Polyclinic EXPERT', Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education Saint Petersburg State University, Clinic of advanced medical technologies n.a. Nicolay I. Pirogov, Saint Petersburg
  - State Budgetary Healthcare Institution "Saratov City Clinical Hospital # 5, Saratov
  - Regional State Budgetary Institution of Health "Clinical Hospital №1", Smolensk
- Saudi Arabia (6):
  - National Guard Hospital Jeddah, Jeddah
  - King Abdulaziz University Hospital, Jeddah
  - Prince Sultan Military Medical City, Riyadh
  - National Guard Hospital Riyadh, Riyadh
  - King Fahad Medical City, Riyadh
  - King Khalid University Hospital, Riyadh
- South Africa (4):
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Wits Clinical Research, Johannesburg, Guauteng
  - EMMED, Pretoria, Guauteng
  - Inspired GI Care, Cape Town, Western Cape
- Spain (5):
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Clínico San Carlos and Instituto de Investigación del Hospital Clínico San Carlos (IdISSC), Madrid
  - Hospital Virgen de la Salud, Toledo
- Turkey (Türkiye) (5):
  - SBÜ. Antalya Eğirim ve Araştırma Hastanesi, Gastroenteroloji, Antalya
  - Marmara Universitesi Pendik Eğitim Araştırma Hastanesi, Gastroenteroloji, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Gastroenteroloji, Izmir
  - Mersin Universitesi Tip Fakultesi, Gastroenteroloji, Mersin
  - Karadeniz Teknik Üniversitesi Tıp Fakütesi Hastanesi Gastroenteroloji, Trabzon
- Ukraine (9):
  - Municipal non-profit enterprise "Kharkiv City Clinical Hospital #2 named after prof. O. O. Shalimov" of Kharkiv City Council, Kharkiv
  - Private Enterprise Private Manufacturing Company "Acinus", Kropyvnytskyi
  - Municipal non-profit enterprise "Kyiv City Clinical Hospital No. 18" of the executive body of the Kyiv City Council (Kyiv City State Administration), Kyiv
  - Comunal NonCommercial Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital", Lviv
  - Municipal non-profit enterprise "Odesa Regional Clinical Hospital of the Odesa Regional Council", Regional Gastroenterological Center, Odesa
  - Ternopil University Hospital, Ternopil
  - Municipal non-profit enterprise "M.I. Pyrogov Vinnytsya Regional Clinical Hospital of the Vinnytsya Regional Council"; National Pirogov Memorial Medical University, Vinnytsya, Vinnytsia
  - Municipal non-profit enterprise "Vinnytsya City Clinical Hospital №1"; National Pirogov Memorial Medical University, Vinnytsya, Vinnytsia
  - Limited Liability Company "Medibor", Zhytomyr
- Vietnam (10):
  - 103 Military Hospital, Hanoi
  - Bach Mai Hospital, Hanoi
  - Hanoi Medical University Hospital, Hanoi
  - Viet Duc Hospital, Hanoi
  - Vinmec Hospital, Hanoi
  - 115 People's Hospital, Ho Chi Minh City
  - Cho Ray Hospital, Ho Chi Minh City
  - Gia Dinh People's Hospital, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City
  - Hue Central Hospital, Huế

IPD SHARING:
Plan to Share IPD: No